CLINICAL TRIAL: NCT05671328
Title: Evaluation of the Incidence of Invasive Pulmonary Aspergillosis in Patients With Suspected Ventilator-associated Pneumonia
Brief Title: Incidence of Invasive Pulmonary Aspergillosis in Ventilator-associated Pneumonia
Acronym: ASPIC
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022_0061; 2022-A00496-37 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2022-12-15; First posted 2023-01-04 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Ventilator Associated Pneumonia; Pulmonary Aspergillosis Invasive
Keywords: Pulmonary invasive aspergillosis; ventilator-associated-pneumonia; mechanical ventilation; nosocomial infections
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Invasive Pulmonary Aspergillosis; Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with suspected ventilator-associated pneumonia
  Interventions: Other: Biological examinations performed on blood and BAL

INTERVENTIONS:
Other: Biological examinations performed on blood and BAL — Direct examination and culture of BAL Galactomannan in serum and BAL Serum 1,3 beta D glucans Aspergillus PCR in BAL

SUMMARY:
Mechanically ventilated patients are at risk of developing ventilator-associated pneumonia (VAP). Invasive pulmonary aspergillosis (IPA), the diagnosis of which motivates the implementation of specific treatments, is one of the causes of VAP. The hypothesis of the study is that the incidence of IPA is 12.4%. For each patient presenting with a suspicion of VAP and requiring a bronchoalveolar lavage (BAL), the diagnosis of API will be evaluated by biological examinations performed on blood and BAL. Medical and surgical history as well as clinical and biological data will be collected for 28 days or until discharge from the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age ≥ 18 years),
* On invasive ventilation for more than 48 hours,
* Suspected VAP, defined by the appearance or worsening of a radiological pulmonary infiltrate, associated with 2 of the following clinical criteria:

  * Fever ≥ 38° C or hypothermia ≤ 36.5° C
  * Leukocytes > 12x109 or < 4x109/L
  * Purulent tracheal secretions

Exclusion Criteria:

* Neutropenic patients (neutrophils < 0.5G/L),
* Previous diagnosis of IPA,
* Minor patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in ICU
Sampling Method: Non-Probability Sample
Enrollment: 263 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
Incidence of probable or proven IPA according to the Verweij criteria in patients with suspected VAP | On the 1 day of inclusion

SECONDARY OUTCOMES:
Incidence of IPA according to the Blot criteria | On the 1 day of inclusion
Incidence of Aspergillus tracheobronchitis associated with IPA according to the Verweij criteria | On the 1 day of inclusion
Incidence of IPA according to the Verweij criteria in the subgroup without risk factors. | On the 1 day of inclusion
Mortality | at 28 days
Length of stay in intensive care unit | Until discharge from the ICU, an average 28 days
Duration of mechanical ventilation | Until discharge from the ICU, an average 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Saad NSEIR, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Pôle de Réanimation Hôpital R. Salengro, CHU de Lille, Lille, France